

## DIRECCIÓN DE PRESTACIONES MÉDICAS

Coordinación de Investigación en Salud División de Innovación y Regulación de la Investigación en Salud Comité de Ética en Investigación

Ciudad de México, a 12 de enero de 2024.

## Dr. José de Jesús Peralta Romero

Investigador Responsable Unidad de Investigación Médica en Bioquímica UMAE, Centro Médico Nacional Siglo XXI Presente

En relación con el protocolo titulado: "EVALUACIÓN DEL EFECTO DE LA ELECTROACUPUNTURA EN LOS SÍNTOMAS SENSITIVOS DE LA POLINEUROPATÍA DISTAL SIMÉTRICA DE ORIGEN DIABÉTICO Y SU CORRELACIÓN CON CAMBIOS EN LA VELOCIDAD DE CONDUCCIÓN NERVIOSA", con número de registro 2020-785-070, el Comité de Ética en Investigación CONBIOÉTICA-09-CEI-009-20160601, revisó y aprobó la solicitud de reaprobación anual del proyecto por el periodo del 10 de enero de 2024 al 9 de enero de 2025. A su vez, se aprueba el cronograma de actualizado.

Sin otro particular, reciba un cordial saludo.

Atentamente

Dra. Marcela Pérez Rodríguez

Presidente Comité de Ética en Investigación Coordinación de Investigación en Salud Centro Médico Nacional Siglo XXI

RBB/mcjbm/ F-CNIC-2019-068

